CLINICAL TRIAL: NCT01169948
Title: 320 Multidetector Computed Tomography in the Preoperative Assessment for Coronary Artery Bypass Graft Surgery
Brief Title: 320 Multidetector Computed Tomography Prior to Coronary Artery Bypass Surgery
Status: Withdrawn | Type: Observational
Why Stopped: Not funded.
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 2009/R/CAR/17
Record Dates: First submitted 2010-07-14; First posted 2010-07-26 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Coronary Disease
Keywords: Coronary disease; Coronary artery bypass; Cardiac surgery; Computed tomography; Coronary angiography
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients awaiting cardiac surgery
  Interventions: Radiation: Computed tomography scan

INTERVENTIONS:
Radiation: Computed tomography scan — Computed tomography will be performed using a 320 multidetector computed tomography scanner and may include coronary calcium score, coronary angiography and myocardial perfusion scanning.

SUMMARY:
Recent advances in technology have resulted in the development of scanners that can n image the heart arteries within 10 to 20 minutes but without the need for admission to hospital or insertion of catheters. This means that coronary heart disease may be more readily identified (or ruled out) and allow better diagnosis and treatment of patients with symptoms suggesting coronary heart disease. Here, we propose to assess the latest and most powerful scanners to see if it can accurately diagnose the extent of coronary artery disease and facilitate the planning of heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients who have undergone conventional coronary angiography and have been referred for coronary artery bypass surgery or valve replacement

Exclusion Criteria:

* age less than 18
* pregnancy or breast feeding
* inability to undergo computed tomography scanning
* inability to give informed consent
* severe renal failure (serum creatinine >250umol/l or estimated glomerular filtration rate <15ml/min)
* known allergy to iodinated contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients awaiting cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-06

PRIMARY OUTCOMES:
Coronary artery stenosis defined qualitatively by trained observers and quantitatively by computer software | 1 month

SECONDARY OUTCOMES:
Myocardial perfusion defects defined qualitatively by trained observers and quantitatively by computer software | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, PhD BM DM, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Scotland, United Kingdom